CLINICAL TRIAL: NCT07343687
Title: Clinico-hematological and Coagulation Profiles in Newly Diagnosed Acute Myeloid Leukemia Patients Treated With Intensive Induction Chemotherapy .
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa Mahmoud Ahmed, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: clinicohematological AML
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Newly diagnosed AML patients (age ≥18) Undergoing intensive induction therapy

SUMMARY:
Acute myeloid leukemia (AML) is a heterogeneous hematological malignancy characterized by clonal proliferation of myeloid precursors in the bone marrow, leading to impaired hematopoiesis and bone marrow failure[1,2]. Which results in ineffective erythropoiesis and megakaryopoiesis , clinically manifesting as relatively rapid bone marrow failure compared to chronic and indolent leukemias. This lead to inadequate production of red blood cells and platelets. Patients with AML frequently present with cytopenias, including thrombocytopenia, which significantly increases the risk of bleeding complications. Bleeding is a major clinical concern in AML, with studies reporting that 40-70% of patients experience bleeding manifestations at diagnosis[3,4].

Disseminated intravascular coagulation is a particularly significant complication in AML, occurring in 10-40% of patients at presentation. The presence of overt DIC at diagnosis has been shown to be a strong predictor of both bleeding and thrombotic events, as well as early mortality in AML patients[7,8]. The pathogenesis of DIC in AML is thought to involve the release of tissue factor-like material and cytokines from leukemic blasts, which activate the coagulation cascade and lead to widespread fibrin formation and consumption of clotting factors. This consumptive coagulopathy results in a paradoxical state where patients are at risk for both thrombosis and severe bleeding[7,8].

In addition to DIC, primary hemostatic defects have been identified as important contributors to bleeding risk in AML. Studies have demonstrated that von Willebrand factor (vWF) activity, specifically vWF ristocetin cofactor activity (vWF:RCo), is significantly reduced in AML patients at diagnosis and correlates with the severity of bleeding manifestations[9,10]. Lower vWF:RCo activity has been observed in patients with major bleeding episodes, suggesting its potential as a prognostic marker for bleeding risk independent of other laboratory parameters. Furthermore, alterations in factor VIII activity and other components of the coagulation cascade have been implicated in the pathogenesis of bleeding in AML[9,10].

Treatment options vary depending on patient-specific factors, and hematopoietic stem cell transplant remains the only curative therapy. Although the administration of multi-agent induction chemotherapy can achieve complete remission , allogeneic stem cell transplantation is the only established curative therapy. Despite advancements in therapeutic approaches, prognosis remains suboptimal , specially among the older populations.[15,16,17].

Laboratory evaluation of coagulation profiles in AML typically includes assessment of prothrombin time (PT), activated partial thromboplastin time (aPTT), fibrinogen levels, and D-dimer, which help to identify and monitor coagulopathy and fibrinolysis. Studies have shown significant differences in PT between acute and chronic leukemia patients, highlighting the importance of coagulation testing in the acute setting. The International Society on Thrombosis and Haemostasis (ISTH) DIC score has emerged as a valuable tool for predicting early mortality and guiding clinical management in AML patients with coagulopathy[11,12].

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML patients (age ≥18).
* Undergoing intensive induction therapy (Idarubicin 12 mg/m2 per day for 2-3 days , and cyarabine 100mg /day For 5-7 days ).

Exclusion Criteria:

* * AML (M3).

  * Relapsed patients with AML.
  * patients with AML who started chemotherapy before enrollment in the study.
  * AML with antecedent hematologic malignancy ,or solid tumors.
  * Abnormal liver function tests, known liver disease.
  * Pregnancy.
  * Chronic kidney disease : moderate to severe stage.
  * Prior anticoagulant use.
  * Active infection/sepsis on admission.
  * DIC from other causes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed AML patients (age ≥18).
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
coagulation profile abnormalities | 3 month
  difference in coagulation profile abnormalities in Newly diagnosed AML patients before and after treatment with intensive Induction chemotherapy.